CLINICAL TRIAL: NCT01564745
Title: Cough Determinants in Mechanically Ventilated Patients: a Physiological Study
Brief Title: Cough Determinants in Mechanically Ventilated Patients
Acronym: Extu-Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Extu-Cough
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2014-02

CONDITIONS: Mechanical Ventilation
MeSH Terms: interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cough Determinants (Other)
  Interventions: Other: Functional respiratory evaluation

INTERVENTIONS:
Other: Functional respiratory evaluation — Each enrolled patients has a pulmonary function test before and after extubation, and repeatedly at D1, D3, D5 (if they are always hospitalized)
  Other Names: Pulmonary Function test

SUMMARY:
In our knowledge there is only few data about the cough determinants in mechanically ventilated patients. However some failure of extubation is due to inefficiency cough. In order to determine some determinants of cough, the investigators propose to evaluate systematically different physiological parameters before and after extubation.

DETAILED DESCRIPTION:
In order to evaluate, and identify the cough determinants, the investigators propose a physiological evaluation for each patients who were intubated and mechanically ventilated during at least 72 hours. Indeed inefficacy of cough after extubation is one of the main reason of extubation failure. However there is no any mean to evaluate it simply now.

ELIGIBILITY:
Inclusion Criteria:

* Patients mechanically ventilated since 72h
* Age > 18 years
* Hospitalized in Intensive care Unit
* In weaning phase - with the classically criteria to be extubated
* Patients who passed the weaning test (T tube test or other)

Exclusion Criteria:

* Hemodynamic instability
* Absence of consent
* No cooperation of the patient
* Hemodynamic instability
* pH < 7,30
* Severe hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Interest of systematically cough evaluation before extubation | 2 days after extubation
  All the patients enrolled have a physiological evaluation before and after extubation. After extubation the evaluation will be done respectively at D0, D1, D3 and D5. The first endpoint is the success of extubation which is evaluated à D2.

SECONDARY OUTCOMES:
Correlation between success of extubation and respiratory parameters | 2 days after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas TERZI, MD - PhD, Principal Investigator — University Hospital, Caen; Frédéric Lofaso, MD-PhD, Principal Investigator — University Hospital, Garches; David Orlikowski, MD-PhD, Principal Investigator — University Hospital, Garches
Locations (2):
- France (2):
  - University Hospital, Caen, Caen
  - University Hospital, Garches, Garches

REFERENCES:
- [Derived] Terzi N, Lofaso F, Masson R, Beuret P, Normand H, Dumanowski E, Falaize L, Sauneuf B, Daubin C, Brunet J, Annane D, Parienti JJ, Orlikowski D. Physiological predictors of respiratory and cough assistance needs after extubation. Ann Intensive Care. 2018 Feb 5;8(1):18. doi: 10.1186/s13613-018-0360-3. PMID 29404723